CLINICAL TRIAL: NCT00591786
Title: A Multi-center, Randomized, Open-label, Prospective Bridging, Parallel Dose Finding Trial Comparing Efficacy and Safety of 5 Doses of Org 25969 Administered at 1-2 PTC After Rocuronium or Vecuronium in Japanese and Caucasian Subjects. Part A: Japanese Subjects.
Brief Title: A Bridging Trial Comparing Sugammadex (Org 25969) at 1-2 Post-Tetanic Count (PTC) in Japanese Participants. Part A (P05957)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05957; 2005-001133-15 (EudraCT Number); MK-8616-031 (Other: Merck Protocol Number); 19.4.209A (Other: Organon Protocol Number)
Record Dates: First submitted 2007-12-27; First posted 2008-01-11 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Sugammadex 0.5 mg/kg (Rocuronium) (Experimental): After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered intravenously (IV), followed by maintenance doses of 0.1-0.2 mg/kg rocuronium IV if necessary. At reappearance of the second twitch (T2) response to Train-of-four (TOF) stimulation, a single dose of 0.5 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex
- Sugammadex 1.0 mg/kg (Rocuronium) (Experimental): After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered IV, followed by maintenance doses of 0.1-0.2 mg/kg rocuronium IV if necessary. At reappearance of the T2 response to TOF stimulation, a single dose of 1.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex
- Sugammadex 2.0 mg/kg (Rocuronium) (Experimental): After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered IV, followed by maintenance doses of 0.1-0.2 mg/kg rocuronium IV if necessary. At reappearance of the T2 response to TOF stimulation, a single dose of 2.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex
- Sugammadex 4.0 mg/kg (Rocuronium) (Experimental): After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered IV, followed by maintenance doses of 0.1-0.2 mg/kg rocuronium IV if necessary. At reappearance of the T2 response to TOF stimulation, a single dose of 4.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex
- Sugammadex 8.0 mg/kg (Rocuronium) (Experimental): After induction of anesthesia an intubation dose of 0.9 mg/kg rocuronium was administered IV, followed by maintenance doses of 0.1-0.2 mg/kg rocuronium IV if necessary. At reappearance of the T2 response to TOF stimulation, a single dose of 0.8 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex
- Sugammadex 0.5 mg/kg (Vecuronium) (Experimental): After induction of anesthesia an intubation dose of 0.1 mg/kg vecuronium was administered IV, followed by maintenance doses of 0.02-0.4 mg/kg vecuronium IV if necessary. At reappearance of the T2 response to TOF stimulation, a single dose of 0.5 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex
- Sugammadex 1.0 mg/kg (Vecuronium) (Experimental): After induction of anesthesia an intubation dose of 0.1 mg/kg vecuronium was administered IV, followed by maintenance doses of 0.02-0.4 mg/kg vecuronium IV if necessary. At reappearance of the T2 response to TOF stimulation, a single dose of 1.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex
- Sugammadex 2.0 mg/kg (Vecuronium) (Experimental): After induction of anesthesia an intubation dose of 0.1 mg/kg vecuronium was administered IV, followed by maintenance doses of 0.02-0.4 mg/kg vecuronium IV if necessary. At reappearance of the T2 response to TOF stimulation, a single dose of 2.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex
- Sugammadex 4.0 mg/kg (Vecuronium) (Experimental): After induction of anesthesia an intubation dose of 0.1 mg/kg vecuronium was administered IV, followed by maintenance doses of 0.02-0.4 mg/kg vecuronium IV if necessary. At reappearance of the T2 response to TOF stimulation, a single dose of 4.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex
- Sugammadex 8.0 mg/kg (Vecuronium) (Experimental): After induction of anesthesia an intubation dose of 0.1 mg/kg vecuronium was administered IV, followed by maintenance doses of 0.02-0.4 mg/kg vecuronium IV if necessary. At reappearance of the T2 response to TOF stimulation, a single dose of 8.0 mg/kg sugammadex was administered IV.
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Sugammadex — After induction of anesthesia an intubation dose of a neuromuscular blocking agent (NMBA) was administered IV: either 0.9 mg/kg rocuronium (arms 1-5) or 0.1 mg/kg vecuronium (arms 6-10). Maintenance doses of 0.1-0.2 mg/kg rocuronium IV or 0.02-0.04 mg/kg vecuronium IV could be administered if necessary. At reappearance of T2 the randomized single dose of sugammadex (0.5 to 8.0 mg/kg) IV was administered.
  Other Names: Org 25969; MK-8616; Bridion®

SUMMARY:
The objective of the trial was to establish the dose-response relation of sugammadex (Org 25969) given as a reversal agent of rocuronium or vecuronium at 1-2 PTC during sevoflurane anesthesia for Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants of American Society of Anesthesiologists (ASA) class 1 - 3;
* Participants at least 20 years but under 65 years of age;
* Japanese participants;
* Participants scheduled for elective surgery in supine position and under sevoflurane anesthesia, in need of administration of a neuromuscular blocking agent (NMBA), with an anticipated duration of about 1.5-3 hours;
* Participants who had given written informed consent. This was obtained before the investigator or the sub-investigator performed any procedures or assessments for the screening, and after the participant was informed about the nature and purpose of the study, the study procedures, and the risks and restrictions of the study.

Exclusion Criteria:

* Participants in whom a difficult intubation because of anatomical malformations was expected;
* Participants known or suspected to have neuromuscular disorders impairing neuromuscular blockade (NMB) and/or significant renal dysfunction (for example a creatinine level > 1.6 mg/dl) and/or severe hepatic dysfunction.
* Participants known or suspected to have a (family) history of malignant hyperthermia;
* Participants known or suspected to have an allergy to narcotics, muscle relaxants or other medication used during general anesthesia;
* Participants receiving medication expected to interfere with the rocuronium or vecuronium given in this trial, based on the dose and time of administration;
* Female participants who were pregnant;
* Female participants of childbearing potential not using birth control or using only oral contraception as birth control;
* Participants who were breast-feeding;
* Participants who had already participated in study CT 19.4.209A, or in another trial with sugammadex;
* Participants who had participated in another clinical trial within 6 months of entering into study CT 19.4.209A.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-12-05 (Actual); Primary Completion 2006-08-31 (Actual); Study Completion 2006-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Takeda J, Iwasaki H, Otagiri T, Katoh T, Shingu K, Obara H, Nakatsuka H, Tomiyama Y, Kasaba T. [Efficacy and safety of sugammadex (Org 25969) in reversing deep neuromuscular block induced by rocuronium or vecuronium in Japanese patients]. Masui. 2014 Oct;63(10):1083-8. Japanese. PMID 25693333
- See also: Click here to access a synopsis of the study results. — http://www.merck.com/clinical-trials/policies-perspectives.html
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugammadex 0.5 mg/kg (Rocuronium): Sugammadex 0.5 mg/kg administered as a single-bolus intravenous (IV) dose at 1-2 Post-tetanic count (PTC) after 0.9 mg/kg rocuronium (single-bolus IV dose) for intubation, followed by maintenance doses of rocuronium 0.1-0.2 mg/kg if necessary
- Sugammadex 1.0 mg/kg (Rocuronium): Sugammadex 1.0 mg/kg administered as a single-bolus IV dose at 1-2 PTC after 0.9 mg/kg rocuronium (single-bolus IV dose) for intubation, followed by maintenance doses of rocuronium 0.1-0.2 mg/kg if necessary
- Sugammadex 2.0 mg/kg (Rocuronium): Sugammadex 2.0 mg/kg administered as a single-bolus IV dose at 1-2 PTC after 0.9 mg/kg rocuronium (single-bolus IV dose) for intubation, followed by maintenance doses of rocuronium 0.1-0.2 mg/kg if necessary
- Sugammadex 4.0 mg/kg (Rocuronium): Sugammadex 4.0 mg/kg administered as a single-bolus IV dose at 1-2 PTC after 0.9 mg/kg rocuronium (single-bolus IV dose) for intubation, followed by maintenance doses of rocuronium 0.1-0.2 mg/kg if necessary
- Sugammadex 8.0 mg/kg (Rocuronium): Sugammadex 8.0 mg/kg administered as a single-bolus IV dose at 1-2 PTC after 0.9 mg/kg rocuronium (single-bolus IV dose) for intubation, followed by maintenance doses of rocuronium 0.1-0.2 mg/kg if necessary
- Sugammadex 0.5 mg/kg (Vecuronium): Sugammadex 0.5 mg/kg administered as a single-bolus IV dose at 1-2 PTC after 0.1 mg/kg vecuronium (single-bolus IV dose) for intubation, followed by maintenance doses of vecuronium 0.02-0.04 mg/kg if necessary
- Sugammadex 1.0 mg/kg (Vecuronium): Sugammadex 1.0 mg/kg administered as a single-bolus IV dose at 1-2 PTC after 0.1 mg/kg vecuronium (single-bolus IV dose) for intubation, followed by maintenance doses of vecuronium 0.02-0.04 mg/kg if necessary
- Sugammadex 2.0 mg/kg (Vecuronium): Sugammadex 2.0 mg/kg administered as a single-bolus IV dose at 1-2 PTC after 0.1 mg/kg vecuronium (single-bolus IV dose) for intubation, followed by maintenance doses of vecuronium 0.02-0.04 mg/kg if necessary
- Sugammadex 4.0 mg/kg (Vecuronium): Sugammadex 4.0 mg/kg administered as a single-bolus IV dose at 1-2 PTC after 0.1 mg/kg vecuronium (single-bolus IV dose) for intubation, followed by maintenance doses of vecuronium 0.02-0.04 mg/kg if necessary
- Sugammadex 8.0 mg/kg (Vecuronium): Sugammadex 8.0 mg/kg administered as a single-bolus IV dose at 1-2 PTC after 0.1 mg/kg vecuronium (single-bolus IV dose) for intubation, followed by maintenance doses of vecuronium 0.02-0.04 mg/kg if necessary
Period: Overall Study
Arm/Group | Sugammadex 0.5 mg/kg (Rocuronium) | Sugammadex 1.0 mg/kg (Rocuronium) | Sugammadex 2.0 mg/kg (Rocuronium) | Sugammadex 4.0 mg/kg (Rocuronium) | Sugammadex 8.0 mg/kg (Rocuronium) | Sugammadex 0.5 mg/kg (Vecuronium) | Sugammadex 1.0 mg/kg (Vecuronium) | Sugammadex 2.0 mg/kg (Vecuronium) | Sugammadex 4.0 mg/kg (Vecuronium) | Sugammadex 8.0 mg/kg (Vecuronium)
Started | 9 | 9 | 11 | 11 | 10 | 10 | 10 | 10 | 10 | 10
Treated Participants | 9 | 9 | 10 | 11 | 10 | 10 | 10 | 10 | 10 | 10
Completed | 9 | 9 | 10 | 11 | 10 | 10 | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal of Informed Consent | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Participants
Groups:
- Sugammadex 2.0 mg/kg (Rcocuronium): Sugammadex 2.0 mg/kg administered as a single-bolus IV dose at 1-2 PTC after 0.9 mg/kg rocuronium (single-bolus IV dose) for intubation, followed by maintenance doses of rocuronium 0.1-0.2 mg/kg if necessary
- Total: Total of all reporting groups
Arm/Group | Sugammadex 0.5 mg/kg (Rocuronium) | Sugammadex 1.0 mg/kg (Rocuronium) | Sugammadex 2.0 mg/kg (Rcocuronium) | Sugammadex 4.0 mg/kg (Rocuronium) | Sugammadex 8.0 mg/kg (Rocuronium) | Sugammadex 0.5 mg/kg (Vecuronium) | Sugammadex 1.0 mg/kg (Vecuronium) | Sugammadex 2.0 mg/kg (Vecuronium) | Sugammadex 4.0 mg/kg (Vecuronium) | Sugammadex 8.0 mg/kg (Vecuronium) | Total
Number analyzed (Participants) | 9 | 9 | 10 | 11 | 10 | 10 | 10 | 10 | 10 | 10 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (13) | 48 (13) | 45 (13) | 48 (13) | 44 (13) | 44 (14) | 51 (10) | 40 (13) | 38 (11) | 50 (12) | 45 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 3 | 3 | 8 | 4 | 3 | 5 | 4 | 5 | 45
  Male | 4 | 4 | 7 | 8 | 2 | 6 | 7 | 5 | 6 | 5 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Japanese: Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Japanese: Not Hispanic or Latino | 9 | 9 | 10 | 11 | 10 | 10 | 10 | 10 | 10 | 10 | 99
  Japanese: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time From Start of Sugammadex Administration to Recovery of the Neuromuscular Response to a Ratio of 0.9 for Train-Of-Four (TOF) Stimulation
Description: Neuromuscular functioning was monitored by applying repetitive Train-Of-Four (TOF) electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the amplitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from neuromuscular blockade (NMB). In this study, twitch responses were recorded until the T4/T1 Ratio reached >= 0.9, the minimum acceptable ratio that indicated recovery from NMB. A faster time to recovery of the T4/T1 Ratio to 0.9 indicates a faster recovery from NMB.
Time Frame: Up to 269:45 (min:sec)
Population: The analysis population consisted of all randomized participants who were given at least one administration of sugammadex and had at least one post-baseline efficacy measurement, without any major protocol violation.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sugammadex 0.5 mg/kg (Rocuronium) | Sugammadex 1.0 mg/kg (Rocuronium) | Sugammadex 2.0 mg/kg (Rocuronium) | Sugammadex 4.0 mg/kg (Rocuronium) | Sugammadex 8.0 mg/kg (Rocuronium) | Sugammadex 0.5 mg/kg (Vecuronium) | Sugammadex 1.0 mg/kg (Vecuronium) | Sugammadex 2.0 mg/kg (Vecuronium) | Sugammadex 4.0 mg/kg (Vecuronium) | Sugammadex 8.0 mg/kg (Vecuronium)
Number analyzed (Participants) | 6 | 7 | 10 | 11 | 10 | 5 | 7 | 10 | 10 | 10
Minutes | 66.90 (34.63) | 4.73 (1.73) | 3.43 (2.52) | 1.58 (0.88) | 1.32 (0.57) | 79.48 (46.23) | 39.82 (45.77) | 16.02 (42.20) | 3.05 (2.38) | 2.93 (3.77)

2. Secondary Outcome: Time From Start of Sugammadex Administration to Recovery of the Neuromuscular Response to a Ratio of 0.7 for TOF Stimulation
Description: Neuromuscular functioning was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the amplitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB. A faster time to recovery of the T4/T1 Ratio to 0.7 indicates a faster recovery from NMB.
Time Frame: Up to 152:30 (min:sec)
Population: The analysis population was the Per-Protocol (PP) group, which consisted of all randomized participants who were given at least one administration of sugammadex and had at least one post-baseline efficacy measurement, without any major protocol violation.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sugammadex 0.5 mg/kg (Rocuronium) | Sugammadex 1.0 mg/kg (Rocuronium) | Sugammadex 2.0 mg/kg (Rocuronium) | Sugammadex 4.0 mg/kg (Rocuronium) | Sugammadex 8.0 mg/kg (Rocuronium) | Sugammadex 0.5 mg/kg (Vecuronium) | Sugammadex 1.0 mg/kg (Vecuronium) | Sugammadex 2.0 mg/kg (Vecuronium) | Sugammadex 4.0 mg/kg (Vecuronium) | Sugammadex 8.0 mg/kg (Vecuronium)
Number analyzed (Participants) | 6 | 9 | 10 | 11 | 10 | 7 | 9 | 10 | 10 | 10
Minutes | 34.45 (32.12) | 4.38 (2.32) | 2.48 (2.00) | 1.07 (0.20) | 1.03 (0.32) | 56.82 (35.47) | 8.30 (10.90) | 3.18 (3.72) | 1.95 (1.35) | 1.33 (0.58)

3. Secondary Outcome: Time From Start of Sugammadex Administration to Recovery of the Neuromuscular Response to a Ratio of 0.8 for TOF Stimulation
Description: Neuromuscular functioning was monitored by applying repetitive TOF electrical stimulations to the ulnar nerve every 15 seconds and assessing twitch response at the adductor pollicis muscle. T1 and T4 refer to the amplitudes (heights) of the first and fourth twitches, respectively, after TOF nerve stimulation. The T4/T1 Ratio (expressed as a decimal of up to 1.0) indicates the extent of recovery from NMB. A faster time to recovery of the T4/T1 Ratio to 0.8 indicates a faster recovery from NMB.
Time Frame: Up to 194:45 (min:sec)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sugammadex 0.5 mg/kg (Rocuronium) | Sugammadex 1.0 mg/kg (Rocuronium) | Sugammadex 2.0 mg/kg (Rocuronium) | Sugammadex 4.0 mg/kg (Rocuronium) | Sugammadex 8.0 mg/kg (Rocuronium) | Sugammadex 0.5 mg/kg (Vecuronium) | Sugammadex 1.0 mg/kg (Vecuronium) | Sugammadex 2.0 mg/kg (Vecuronium) | Sugammadex 4.0 mg/kg (Vecuronium) | Sugammadex 8.0 mg/kg (Vecuronium)
Number analyzed (Participants) | 6 | 8 | 10 | 11 | 10 | 6 | 8 | 10 | 10 | 10
Minutes | 46.78 (30.85) | 4.33 (1.85) | 2.98 (2.17) | 1.33 (0.58) | 1.13 (0.40) | 73.25 (45.65) | 22.60 (27.90) | 6.02 (11.83) | 2.22 (1.48) | 1.42 (0.53)

ADVERSE EVENTS:
Time Frame: Up to 7 post-operative days
Description: All randomized participants who received at least one dose of study treatment and had follow-up.
Arm/Group | Sugammadex 0.5 mg/kg (Rocuronium) | Sugammadex 1.0 mg/kg (Rocuronium) | Sugammadex 2.0 mg/kg (Rocuronium) | Sugammadex 4.0 mg/kg (Rocuronium) | Sugammadex 8.0 mg/kg (Rocuronium) | Sugammadex 0.5 mg/kg (Vecuronium) | Sugammadex 1.0 mg/kg (Vecuronium) | Sugammadex 2.0 mg/kg (Vecuronium) | Sugammadex 4.0 mg/kg (Vecuronium) | Sugammadex 8.0 mg/kg (Vecuronium)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/10 | 0/11 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/9 | 0/10 | 0/11 | 0/10 | 0/10 | 0/10 | 1/10 | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 9/9 | 9/9 | 10/10 | 11/11 | 10/10 | 10/10 | 9/10 | 10/10 | 9/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex 0.5 mg/kg (Rocuronium) (N=9) | Sugammadex 1.0 mg/kg (Rocuronium) (N=9) | Sugammadex 2.0 mg/kg (Rocuronium) (N=10) | Sugammadex 4.0 mg/kg (Rocuronium) (N=11) | Sugammadex 8.0 mg/kg (Rocuronium) (N=10) | Sugammadex 0.5 mg/kg (Vecuronium) (N=10) | Sugammadex 1.0 mg/kg (Vecuronium) (N=10) | Sugammadex 2.0 mg/kg (Vecuronium) (N=10) | Sugammadex 4.0 mg/kg (Vecuronium) (N=10) | Sugammadex 8.0 mg/kg (Vecuronium) (N=10)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex 0.5 mg/kg (Rocuronium) (N=9) | Sugammadex 1.0 mg/kg (Rocuronium) (N=9) | Sugammadex 2.0 mg/kg (Rocuronium) (N=10) | Sugammadex 4.0 mg/kg (Rocuronium) (N=11) | Sugammadex 8.0 mg/kg (Rocuronium) (N=10) | Sugammadex 0.5 mg/kg (Vecuronium) (N=10) | Sugammadex 1.0 mg/kg (Vecuronium) (N=10) | Sugammadex 2.0 mg/kg (Vecuronium) (N=10) | Sugammadex 4.0 mg/kg (Vecuronium) (N=10) | Sugammadex 8.0 mg/kg (Vecuronium) (N=10)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 | 1 (1) | 3 (3) | 0 | 2 (2) | 0 | 2 (2) | 0
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 | 0 | 2 (2) | 2 (2) | 1 (1) | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 0 | 2 (2) | 0 | 1 (1) | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (5) | 3 (3) | 2 (2) | 5 (6) | 2 (2) | 4 (4) | 2 (2) | 4 (4) | 3 (3)
Palatal oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1)
Stomach discomfort (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 1 (1) | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 | 0 | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Chills (General disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 1 (1)
Injection site pruritus (General disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 1 (1) | 0
Oedema peripheral (General disorders) | 0 | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 | 0 | 0 | 0 | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) | 0 | 0 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 (1) | 1 (1) | 0 | 2 (2) | 1 (1) | 1 (1) | 0 | 0 | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) | 1 (1) | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 2 | 0 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (5) | 3 (4) | 1 (1) | 2 (2) | 1 (1) | 0 | 2 (2) | 1 (1)
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 1 (1) | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 8 (8) | 8 (9) | 8 (8) | 10 (10) | 8 (8) | 7 (7) | 7 (7) | 7 (7) | 6 (7) | 7 (7)
Albumin urine present (Investigations) | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 1 (1) | 0
Beta 2 microglobulin urine increased (Investigations) | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (1) | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Dizziness (Nervous system disorders) | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 0 | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 | 0 | 2 (2) | 0 | 0
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 1 (1) | 1 (1) | 0 | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 0 | 2 (2) | 1 (1) | 0 | 0 | 0 | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 1 (1) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0 | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0 | 0 | 2 (2) | 1 (1) | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Corneal oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Application site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling abnormal (General disorders) | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Beta 2 microglobulin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Intraocular pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Pharyngolaryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 (1) | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth socket haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral coldness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 1 (1)
Pyrexia (General disorders) | 3 (3) | 2 (2) | 3 (3) | 4 (4) | 3 (3) | 3 (3) | 2 (2) | 4 (4) | 5 (5) | 1 (1)
Thirst (General disorders) | 0 | 0 | 0 | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint warmth (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeltal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any scientific paper, presentation, or other communication concerning the clinical trial described in the protocol will first be submitted to Sponsor, at least six weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.